CLINICAL TRIAL: NCT02708472
Title: Safety and Efficacy of Synchronized Transcranial Magnetic Stimulation (sTMS) for the Treatment of Generalized Anxiety Disorder (GAD) -An Open Label Investigator Initiated Trial
Brief Title: Safety and Efficacy of Synchronized Transcranial Magnetic Stimulation for the Treatment of Generalized Anxiety Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study never moved forward due to funding constraints.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Wave Neuroscience (Industry)
Responsible Party: Principal Investigator, Mustafa Husain, Vice Chair, Department of Psychiatry, Professor of Psychiatry, Neurology & Medicine, Director, Neuromodulation Research & Therapeutics Program, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 112015-078
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Generalized Anxiety Disorder (GAD)
Keywords: Generalized Anxiety Disorder; synchronized Transcranial Magnetic Stimulation; Anxiety; Neurostimulation; TMS
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label (Experimental): Subjects who qualify will receive daily active synchronized Transcranial Magnetic Stimulation (sTMS) treatments. Treatment will be initiated on Day 1 of the study. Subjects will come to the clinic for 5 daily treatment sessions for a total of 4 treatment weeks (20 treatment sessions). Treatment will be discontinued at the end of Week 4. Subjects will be clinically evaluated for safety and efficacy at the end of each of the four weekly treatment courses.
  At the end of Week 4, subjects who have not met the endpoint of 50% reduction in Hamilton Anxiety Rating Scale (HAM-A) score will be eligible to be considered for 2 additional weeks of daily treatment in an extended phase (for a total of 30 treatment sessions).
  Interventions: Device: synchronized Transcranial Magnetic Stimulation (sTMS)

INTERVENTIONS:
Device: synchronized Transcranial Magnetic Stimulation (sTMS) — Subjects who qualify will receive daily active sTMS treatments with the NeoSync, Inc sTMS device. The device includes an EEG recording module and the device uses a proprietary algorithm to determine the individualized alpha frequency (IAF). The IAF obtained during this baseline recording is used throughout the study.
  The device contains three magnets in the sagittal line above the subject's scalp, which rotate along a transverse axis. sTMS stimulation is delivered broadly over the prefrontal and frontal regions of the brain. These magnets rotate to generate a sinusoidal magnetic field set at precisely the average individualized alpha frequency (IAF). Each therapy session lasts 30 minutes.

SUMMARY:
This clinical trial is an investigator-initiated open label study designed to evaluate the safety and efficacy of sTMS in subjects with Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
Subjects will receive 5 daily treatments per treatment week for 4 weeks (20 treatments). Patients who do not meet a 50% reduction of Hamilton Anxiety Rating Scale (HAM-A) score (non-responders) at 4 weeks will be offered 2 additional treatment weeks for up to 30 treatments total.

Subjects who qualify for enrollment will be followed and assessed using the: Mini International Neuropsychiatric Interview (MINI) for Axis 1, Montreal Cognitive Assessment (MoCA), Hamilton Anxiety Rating Scale (HAM-A), Hamilton Depression Rating Scale (HAM-D17), Generalized Anxiety Disorder 7-item (GAD-7), and Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR16) patient reported scale. Treatment will be initiated on Day 1 of the study and will be continued for a minimum of 4 and a maximum of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects will be 18 - 65 years of age.
2. Primary Diagnosis of Generalized Anxiety Disorder (GAD) confirmed by structured interview using the Mini International Neuropsychiatric Interview (MINI), version 7, with minimum duration of current episode of 3 months
3. Baseline Hamilton Anxiety (HAM-A) score equal or greater than 18
4. The baseline EEG is of sufficient duration and quality that it can be processed for quantitative analysis.
5. Taking less than or equal to 2 psychotropic medications at a stable dose for a minimum of 2 weeks to remain unchanged throughout duration of study.
6. Subjects are willing and able to adhere to the intensive treatment schedule and all required study visits.

Exclusion Criteria:

1. Subjects are unable or unwilling to give informed consent.
2. Primary Diagnosis with the following conditions confirmed by MINI (current unless otherwise stated):

   1. GAD secondary to a general medical condition, or substance-induced.
   2. History of substance abuse or dependence within the past 6 months (except nicotine and caffeine).
   3. Major depressive disorder, bipolar disorder or psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes.
   4. Eating disorder (current or within the past year).
   5. Obsessive compulsive disorder (lifetime).
   6. Post-traumatic stress disorder (current or within the past year).
   7. Attention Deficit Hyperactivity Disorder (ADHD) currently being treated.
3. Subjects meeting criteria for Axis II cluster A or B diagnosis based upon Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria, which in the judgment of the Investigator may hinder the subjects in completing the procedures required by the study protocol.
4. Subjects with a clinically defined neurological disorder including, but not limited to:

   1. Any condition likely to be associated with increased intracranial pressure.
   2. Space occupying brain lesion.
   3. Any history of seizure EXCEPT those therapeutically induced by Electroconvulsive Therapy (ECT). Childhood febrile seizures are acceptable and these subjects may be included in the study.
   4. History of stroke.
   5. Transient ischemic attack within two years.
   6. Cerebral aneurysm.
   7. Dementia (Montreal Cognition Assessment score less than 23).
   8. Parkinson's disease.
   9. Huntington's disease.
   10. Multiple sclerosis.
   11. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold.
5. Subjects with any of the following treatment histories:

   1. TMS within 4 weeks prior to the screening visit or any prior treatment with sTMS
   2. ECT treatment within 1 year prior to the screening visit.
   3. Failure to respond to TMS or ECT treatment (i.e., consistent with Antidepressant Treatment History Form confidence level 3 or higher) in this or any previous episode.
   4. Lifetime history of treatment with Deep Brain Stimulation (DBS) or Vagus Nerve Stimulation (VNS).
   5. Use of any investigational drug or device within 6 months of the screening visit.
6. Subjects are adequately benefiting from current antianxiety medication(s)
7. Significant acute suicide risk as judged by the investigator
8. Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
9. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed.
10. Clinically significant abnormality or clinically significant unstable medical condition, as indicated by medical history, physical examination, ECG results, or clinical laboratory testing, that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results, e.g., any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning.
11. Women who are currently pregnant or not using a medically acceptable means of birth control and women who are breastfeeding.
12. Positive urine drug screen for illicit substances. (A positive urine drug screen at screening may be repeated once prior to randomization).
13. Any condition which in the judgment of the Investigator would prevent the subject from completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-01 (Estimated); Primary Completion 2017-04-01 (Estimated); Study Completion 2018-01-22 (Estimated)

PRIMARY OUTCOMES:
Mean change in score on the Hamilton Anxiety Rating Scale (HAM-A) | Baseline to Week 4

SECONDARY OUTCOMES:
Clinical response on the Hamilton Anxiety Rating Scale | Baseline to Week 4
  Clinical response defined as greater than or equal to 50% reduction of assessment score
Clinical response on the Generalized Anxiety Disorder 7-item scale (GAD-7) | Baseline to Week 4
  Clinical response defined as greater than or equal to 50% reduction of assessment score
Clinical response on the Hamilton Depression Rating Scale (HAM-D17) | Baseline to Week 4
  Clinical response defined as greater than or equal to 50% reduction of assessment score
Clinical response on the Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR16) | Baseline to Week 4
  Clinical response defined as greater than or equal to 50% reduction of assessment score

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa M. Husain, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Ahmad Raza, M.D., Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No